CLINICAL TRIAL: NCT06593691
Title: Examining the Effectiveness of Multiwave Locked System Laser Treatment in Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/09-36
Record Dates: First submitted 2024-07-31; First posted 2024-09-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment group (Active Comparator): In conventional treatment, Hot Pack, TENS, therapeutic ultrasound and exercise program will be given by the hospital staff.
  Interventions: Other: conventional treatment
- Conventional treatment + Multiwave Locked System Laser treatment group (Experimental): Multiwave-locked system laser treatment will be applied by the hospital staff to the group in addition to conventional treatment.
  Interventions: Other: conventional treatment; Other: Conventional treatment + multi-wave locked system laser treatment

INTERVENTIONS:
Other: conventional treatment — Hot Pack, TENS, therapeutic ultrasound, and exercise
Other: Conventional treatment + multi-wave locked system laser treatment — Hot Pack, TENS, therapeutic ultrasound, and exercise + multi-wave locked system laser treatment
  Arms: Conventional treatment + Multiwave Locked System Laser treatment group

SUMMARY:
Patients who come to Tavşanlı Assoc. Prof. Dr. Mustafa Kalemli State Hospital, Physical Therapy, and Rehabilitation Department who have been diagnosed with Chronic Low Back Pain by a physician will be included. Patients will be divided into two groups by the physician: conservative treatment and patients whose treatment program is determined as multi-wave locked system laser treatment in addition to conservative treatment. Pain intensity will be measured with a numerical pain rating scale. The Roland-Morris disability questionnaire will be used to evaluate the functionality of the participants, and the esthesiometer will be used to assess tactile acuity. Pressure pain threshold will be evaluated with the MicroFET 2 device. The Turkish Form of the SF-12 Quality of Life Scale will be used to assess the participants' quality of life. Pittsburgh's sleep quality index will be used to evaluate sleep quality. Patient satisfaction will be evaluated with a numerical rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Volunteering to participate in the study
* Having low back pain that has persisted for at least 3 months

Exclusion Criteria:

* History of surgery in the waist area
* Discopathy at a different level of the spine (Modic Type 3)
* Presence of tumor in the spine
* Infection in the discs
* Having an inflammatory disease
* Presence of neurological involvement
* Fracture
* Spondylosis
* Spinal Stenosis
* Spondylolisthesis
* Radiculopathy
* Having received treatment for low back pain in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
pain intensity | Through study completion, an average of 1 year
  Numerical Pain Rating Scale: Ratings from 0 to 10 range from no pain to the highest pain level imaginable. Studies show that a 2-point change in the evaluation made with this scale indicates a clinically significant change beyond the limits of measurement error.Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.

SECONDARY OUTCOMES:
Functionality | Through study completion, an average of 1 year
  The Roland-Morris Disability Questionnaire: This survey contains 24 questions about the impact of low back pain on a person's functionality. The yes answer given by the people is evaluated as 1 point, the no answer is evaluated as 0 points, and a total score between 0 and 24 is received.The score ranges from 0 (no disability) to 24 (max. disability) depending on the questionnaire used.
Tactile Acuity | Through study completion, an average of 1 year
  Esthesiometer: Measurements will be taken by moving horizontally from the midline where the spinous process of the 3rd lumbar vertebra is located to the dominant part of the person. The evaluation will start from the position where the distance between two points is 0 mm, and the distance will be increased until the person can distinguish between two points. Around this determined threshold, 5 increasing and decreasing evaluations will be made and the average of the evaluation will be taken.
Pressure Pain Thereshold | Through study completion, an average of 1 year
  MicroFET 2: Measurements will be taken 5 centimeters to the right and left of the spinous processes of the 3rd and 5th Lumbal vertebrae, which will be marked before. Two more points (on the tibialis anterior muscle of the right and left legs, 5 centimeters lateral to the tuberosity tibia) will be marked and used for control. The probe will be applied perpendicular to the skin, and the pressure will be gradually increased, starting from the point where no pressure is applied at first. At the point when the feeling of pressure turns into pain, participants will be instructed to call this point. This value will be recorded during the application, and after waiting the required time, additional measurements will be taken to calculate the pressure pain threshold.
Assessment of Quality of life | Through study completion, an average of 1 year
  SF 12: The SF-12 health survey is a self-reported outcome measure designed for use among the general population. It is a 12-item short-form health survey that assesses the same eight health domains as the SF-36 Health Survey. Each health domain score contributes to the Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
Sleep Quality | Through study completion, an average of 1 year
  Pittsburgh Sleep Quality Index: 19 out of 24 questions are self-answered questions. While other questions include questions to get information from a roommate or bed partner, some questions in the index are included in the scoring. There are 7 components and the total score varies between 0 and 21. If the total PSQI score is below 5, sleep quality is considered good, and if it is above 5, sleep quality is considered poor.
Patient Satisfaction | Through study completion, an average of 1 year
  Numerical Rating Scale: Participants will score their satisfaction between 0 and 10, with higher scores indicating a higher level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Işıntaş, Study Director — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No